CLINICAL TRIAL: NCT01563250
Title: Improving the Management of Acute Coronary Syndromes in the Emergency Department Using a Rapid Acute Cardiac Evaluation Pathway
Brief Title: Improving the Management of Acute Coronary Syndromes in the Emergency Department
Acronym: RACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Integrated Medical Research LLC (Other)
Collaborators: Alere San Diego (Industry); New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Robert Birkhahn, MD, Director, Integrated Medical Research LLC
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IMR-001
Record Dates: First submitted 2011-06-09; First posted 2012-03-26 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Cardiac Biomarkers; point of care testing
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Core Laboratory (No Intervention): Patients receiving serial routinely available cardiac biomarker testing in a core laboratory setting using Troponin T. (Roche Centaur)
- Point of Care (Active Comparator): Patients will receive the Point of Care testing intervention using serial cardiac biomarker testing at the bedside including myoglobin, Troponin I and CK-MB. (Triage Cardiac Panel, Alere)
  Interventions: Device: Point of Care testing

INTERVENTIONS:
Device: Point of Care testing — The investigators will implement 6 months of randomized testing periods, 2 weeks each. During this 2 week block, cardiac biomarkers will be tested at the bedside in the ED using the Triage Cardiac Panel that will test for CK-MB, Myoglobin, and Troponin I.
  Each blood sample that is take for point of care testing will be saved. The plasma from the saved sample will be frozen and the sample will be sent to an off-site testing center for high sensitivity troponin testing.
  All patients will be followed at the 30-day mark and those patients who are discharged home from the ED will be followed within 48 hours as well.
  Other Names: Triage Cardiac Panel by Alere
  Arms: Point of Care

SUMMARY:
By using a Rapid Cardiac Evaluation (RACE) pathway in the Emergency Department (ED), the investigators can effectively reduce ED wait times and ED length of stay by decreasing overall hospital admissions and telemetry admissions. In addition, the investigators hypothesize a decrease in mortality of those patients admitted for cardiac evaluation by increasing the patient to health care provider ratio.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of chest pain
* 35 years old or greater

Exclusion Criteria:

* ST elevation MI
* New Left Bundle Branch Block
* Admission regardless of test result
* Leaving ED against medical advice

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
ED length of stay | Average of 3 hours stay in the Emergency Department
  From patient check-in time to patient admit or discharge time

SECONDARY OUTCOMES:
Mortality rate of admitted patients | During hospital admission and at 30 days
  Average hospital stay 3 days.
Hospital Admission Rate | Baseline
  Observing the rate at which physicians admit patients to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany A Byrd, D.O., Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States

REFERENCES:
- [Background] Birkhahn RH, Haines E, Wen W, Reddy L, Briggs WM, Datillo PA. Estimating the clinical impact of bringing a multimarker cardiac panel to the bedside in the ED. Am J Emerg Med. 2011 Mar;29(3):304-8. doi: 10.1016/j.ajem.2009.12.007. Epub 2010 Apr 2. PMID 20825823